CLINICAL TRIAL: NCT04584931
Title: Treatment of Gingival Recession Using Gingival Composite Restoration Versus Coronally Advanced Flap: Controlled Clinical Trial
Brief Title: Treatment of Gingival Recession Using Gingival Composite Restoration Versus Coronally Advanced Flap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed AbdelRaouf Hussein, Lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1:3:7
Record Dates: First submitted 2020-10-03; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of gingival recession with colored composite (Experimental): Composite restoration will be applied to the gingival recession defect
  Interventions: Procedure: restorative intervention
- Treatment of gingival recession with coronally advanced flap (Active Comparator): coronally advanced flap at the gingival defect
  Interventions: Procedure: coronally advanced flap

INTERVENTIONS:
Procedure: coronally advanced flap — flap surgery to achieve root coverage at gingival recession defect
  Arms: Treatment of gingival recession with coronally advanced flap
Procedure: restorative intervention — colored composite restoration to camouflage the gingival recession defect
  Arms: Treatment of gingival recession with colored composite

SUMMARY:
Treatment of gingival recession requires favourable anatomical conditions and the use of invasive surgical approaches. Hence, these procedures are not always indicated in all cases and can cause great pain and morbidity. Coloured composite restorations that mimic the lost gingival tissues can provide a non-invasive and simple solution regardless of the recession soft and hard-tissue conditions.

DETAILED DESCRIPTION:
Gingival recession (also known as marginal tissue recession) is defined as the downward displacement of the soft tissues around teeth that would have been otherwise covering the cemento-enamel junction (CEJ), thus exposing the root surface clinically. Recession is one of the most prevalent mucogingival conditions worldwide, affecting between 30% to 100% of the overall population, and its incidence increases with age. Main concerns regarding recession ranging from unacceptable esthetics to the patient, dentinal hypersensitivity, development of carious and non-carious cervical lesions, or impairment of adequate plaque control.

The ultimate aim for treating gingival recession is to provide complete coverage of the root with optimal esthetics and function. A wide range of surgical interventions have been investigated to provide for successful root coverage including rotational and advanced pedicle flaps, free gingival grafts, or regenerative modalities such as guided tissue regeneration. The predictability of surgical techniques depends on patient related factors such as smoking, oral hygiene care and compliance, defect related conditions like depth, width, gingival thickness and interdental attachment level, and finally, operator related skills and experience.

Coronally advanced flap (CAF) with or without the use of connective tissue graft is considered the gold standard for root coverage due to its ability to achieve complete root coverage in favorable defects, superior esthetic outcomes and blending with surrounding gingiva, and the possible realignment and increase in keratinized tissue height. On the other hand, CAF is faced with multiple drawbacks. Complete root coverage in CAF procedures is not predictable in cases with interdental attachment loss. The surgery poses added morbidity, discomfort and pain, and donor site (if present) may augment these complications. Scar formation as a result of incisions or sutures may reduce the overall esthetic appeal. It requires frequent follow-up visits and arduous post-operative instructions. Post-operative results are not stable over long period of time with frequent relapse. The procedure cannot be performed in cases with systemic contraindications for surgical interventions. And finally, it is time-consuming and requires surgical skill and training of the operator.

To overcome all of the abovementioned drawbacks of CAF, composite resin restorative material with pink shades known as "gingival composite" has been proposed to manage gingival recessions. Root coverage with composite is known to effectively reduce dentinal hypersensitivity effectively. Hence, managing gingival recession with this restorative procedure, the patients concerns regarding esthetics or hypersensitivity can be directly addressed using a simple and fast technique. Compared to CAF, restorative procedure shows less pain, morbidity and bleeding, and it does not involve surgical incisions/sutures and hence avoids no scar formation. Pink composite can be presented as a solution in cases that are not expected to benefit from CAF such as RT3, and it can treat carious and non-carious cervical lesions in one step. In addition, it requires less operative time and can be performed by general practitioners and with conventional armamentarium.

ELIGIBILITY:
Inclusion Criteria:

* participants with at least one buccal gingival recession
* O'Leary plaque index less than 20%
* motivated participants willing to complete the follow up

Exclusion Criteria:

* prior surgical or restorative interventions at the recession defect
* smokers
* pregnant participants
* systemic conditions contraindicating dental management

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
post-operative pain | 7 days
  self-reported pain on visual analogue scale (VAS)

SECONDARY OUTCOMES:
post-operative pain | 1,3,5,14 days
  self-reported pain on VAS
overall quality of life: questionnaire | 6 months
  self reported through a questionnaire
Reported post-operative satisfaction | 6 months
  questionnaire
mean root coverage | 6 months
  percentage
complete root coverage | 6 months
  percentage
Probing depth | baseline, 6 months
  in mm
Recession depth | baseline, 6 months
  in mm
Plaque index | baseline, 6 months
  percentage
Bleeding index | baseline, 6 months
  percentage

IPD SHARING:
Plan to Share IPD: No